CLINICAL TRIAL: NCT05077059
Title: Prevalence of Obesity and Overweight in Primary School Children in the Rhein-Neckar Region in Germany - a Cross-Sectional Study / Adipositasprävalenz Bei Grundschulkindern in Der Rhein-Neckar Region - Eine Querschnittsstudie
Brief Title: Prevalence of Obesity and Overweight in Primary School Children in the Rhein-Neckar Region in Germany
Status: Completed | Type: Observational
Sponsor: Adipositasnetzwerk Rhein-Neckar e.V. (Other)
Collaborators: Gesundheitsamt Heidelberg (Unknown); starScience GmbH (Unknown); Oatly AB (Unknown)
Responsible Party: Sponsor
Other Study IDs: Schools Obesity and Overweight
Record Dates: First submitted 2021-09-21; First posted 2021-10-13 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Overweight, Childhood; Obesity, Childhood; Child Development; Overweight and Obesity; Underweight
Keywords: overweight; obesity; children; cognitive function; cognitive function and weight status
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Thinness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will determine the weight status in primary school children in the Rhein-Neckar Region in Germany and will analyse the development of height and weight in these children during the time of COVID-19 related restrictions by asking parents to provide data from childhood examinations. Additionally, interactions between cognitive abilities and weight-status will be studied.

DETAILED DESCRIPTION:
The prevalence of obesity and overweight is increasing among both adults and children. School and kindergarten closings during the COVID-19 epidemic may have had an additional negative impact on the weight development of the affected children. This study aims to examine the post-lockdown prevalence of overweight and obesity in school children in the second grade in the Rhein-Neckar Region in Germany and look at possible lockdown effects. Additionally, interactions between cognitive abilities and weight-status will be studied.

Anthropometric measurements, interviews as well as cognitive testing will be performed in schools in the summer of 2021 in children in the first grade (class 2020/2021). Parents will be asked to provide measurements from U-childhood-examinations and complete a 3-day food record. The local health authority (Gesundheitsamt) will assist in making a representative selection of schools from different socioeconomic areas and provide data from the pre-school examinations. Collected data will be analyzed and compared to national and international surveys, evaluating the trends of the children's height and weight development. Weight status will be assessed by calculating z-BMI standardized for age and compared with national and international growth charts using both national and WHO classification. Potential interrelation between weight-status, weight development with cognitive performance will be explored.

The study will be able to deliver valuable insights in regards to the health of school children in the Rhein-Neckar Region as well as evaluate the effect of COVID-19 related lockdowns on their health.

ELIGIBILITY:
Inclusion Criteria:

* Written consent from parents and or guardians

Exclusion Criteria:

* Missing consent of parents or guardians

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in the second grade
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
BMI | Between October 2021 and January 2022
  Overweight and obesity will be assessed based on the BMI of the children.
zBMI | Through study completion, an average of 4 months
  zBMI will be calculated using German and WHO growth curves / distributions for evaluating child weight status.

SECONDARY OUTCOMES:
Body weight in kg | Between October 2021 and January 2022
  Body weight in kg during the study visit at schools
Height in cm | Between October 2021 and January 2022
  Height in cm during the study visit at schools
abdominal circumference in cm | Between October 2021 and January 2022
  abdominal circumference in cm during the study visit at schools
Upper arm circumference in cm | Between October 2021 and January 2022
  Upper arm circumference in cm during the study visit at schools
Body weight at the time of the U8 physical examination | Between October 2021 and January 2022
  U-Examinations are standard physical examinations available to all children in Germany at pre-specified timepoints. The results of these is recorded in special booklets, kept by the parents.
Height at the time of the U8 physical examination | Between October 2021 and January 2022
  U-Examinations are standard physical examinations available to all children in Germany at pre-specified timepoints. The results of these is recorded in special booklets, kept by the parents.
BMI at the time of the U8 physical examination | Between October 2021 and January 2022
  U-Examinations are standard physical examinations available to all children in Germany at pre-specified timepoints. The results of these is recorded in special booklets, kept by the parents.
Body weight at the time of the U9 physical examination | Between October 2021 and January 2022
  U-Examinations are standard physical examinations available to all children in Germany at pre-specified timepoints. The results of these is recorded in special booklets, kept by the parents.
Height at the time of the U9 physical examination | Between October 2021 and January 2022
  U-Examinations are standard physical examinations available to all children in Germany at pre-specified timepoints. The results of these is recorded in special booklets, kept by the parents.
BMI at the time of the U9 physical examination | Between October 2021 and January 2022
  U-Examinations are standard physical examinations available to all children in Germany at pre-specified timepoints. The results of these is recorded in special booklets, kept by the parents.
Body weight S1 examination data | Between October 2021 and January 2022
  The S1 examination is an examination performed by the health authorities before a child starts goinig to a school. The records are kept by the health authorities.
Height at the time of the S1 examination data | Between October 2021 and January 2022
  The S1 examination is an examination performed by the health authorities before a child starts goinig to a school. The records are kept by the health authorities.
BMI at the time of the S1 examination data | Between October 2021 and January 2022
  The S1 examination is an examination performed by the health authorities before a child starts goinig to a school. The records are kept by the health authorities.
Eating habits | Between October 2021 and January 2022
  Eating habits will be evaluated using a 3-day food record and a questionnaire
Physical activity | Between October 2021 and January 2022
  Physical activity will be assessed using a modified PAQ-C questionnaire as well as a questionnaire for parents
Cognitive testing: Distractibility | Between October 2021 and January 2022
  Distractibility will be studied by a computer-based test from the KiTAP test battery developed by PSYTEST Psychologische Testsysteme, Herzogenrath, which will be administered to the children.
Cognitive testing: Cognitive flexibility | Between October 2021 and January 2022
  Cognitive flexibility will be studied by a computer-based test from the KiTAP test battery developed by PSYTEST Psychologische Testsysteme, Herzogenrath, which will be administered to the children.
Cognitive testing: Alertness and reactions to multiple stimuli | Between October 2021 and January 2022
  Alertness and reactions to multiple stimuli will be studied by a computer-based test from the KiTAP test battery developed by PSYTEST Psychologische Testsysteme, Herzogenrath, which will be administered to the children.

CONTACTS AND LOCATIONS:
Overall Officials: Erhard Siegel, MD, Principal Investigator — Adipositasnetzwerk Rhein-Neckar
Locations (1):
- Adipositasnetzwerk Rhein-Neckar e.V., Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Samigullin A, Gahlert J, Gross G, Morcos M, Schwertz R, Oste R, Siegel E, Humpert P. A central role of nutrition in cognitive function among primary school children: a cross-sectional analysis. BMC Nutr. 2025 Feb 10;11(1):35. doi: 10.1186/s40795-025-01016-2. PMID 39930520
- [Derived] Samigullin A, Gross G, Gahlert J, Buchenberger S, Morcos M, Schwertz R, Oste R, Siegel E, Humpert P. Impact of Covid-19 lockdowns on the anthropometric development in primary school children in the Rhein-Neckar Region, Germany. BMC Nutr. 2024 May 29;10(1):78. doi: 10.1186/s40795-024-00886-2. PMID 38811974